CLINICAL TRIAL: NCT00945594
Title: Randomized Trial Comparing Outpatient Flexible to Rigid Cystoscopy in Females
Brief Title: Trial Comparing Outpatient Flexible to Rigid Cystoscopy in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Cystoscopy
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Pain
Keywords: flexible cystoscopy; rigid cystoscopy; bladder; outcome assessment; pain measurement
MeSH Terms: conditions — Pain | interventions — Cystoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flexible cystoscopy (Experimental): 16F flexible cysto urethroscope (Storz, Culver city, CA)
  Interventions: Device: Cystoscopy
- Rigid cystoscopy (Experimental): 17F, 70° scope (Storz, Culver city, CA)
  Interventions: Device: Cystoscopy

INTERVENTIONS:
Device: Cystoscopy — A 16 F flexible cysto urethroscope (Storz, Culver city, CA) is used for flexible cystoscopy. When rigid cystoscopy is performed, a 17F, 70° scope (Storz, Culver city, CA)

SUMMARY:
The primary purpose of this study to assess patient pain scores comparing rigid to flexible cystoscopy in females; to assess post procedural complications, including frequency, urgency, infection and time to resolution of these symptoms between the two procedures; to assess physician perception of patient pain or discomfort with flexible or rigid cystoscopy.

DETAILED DESCRIPTION:
This will be a prospective randomized trial study in order to determine to compare rigid and flexible cystoscopy in female patients. Patients will be recruited from OU Physicians Pelvic and Bladder Health clinic. Patients receive an information leaflet describing the procedure prior to their appointment. All procedures are performed by the attending physician. Procedures performed by residents and/or fellows are excluded from this study. The vulva is cleaned with antiseptic solution and 10 ml of Xylocaine 2% is be instilled into the urethra before the endoscope was introduced. A 16 F flexible cysto urethroscope (Storz, Culver city, CA) is used for flexible cystoscopy. When rigid cystoscopy is performed, a 17F, 70° scope (Storz, Culver city, CA) is used to enable optimal visualization of the lateral bladder wall in those with previous continence surgeries. The investigator may choose to use a 30° scope when appropriate. Cystoscopy is commenced by recording a postvoid residual ensuring appropriate bladder emptying prior to filling. Filling is performed with continuous saline infusion until the maximum tolerated capacity or 300 ml. (whichever was reached first). A standard systematic approach was adopted to ensure global assessment of the vesical surface. This included the bladder dome, the bladder neck, bladder trigone, sidewalls and ureteral orifices. The urethroscopy portion of the procedure is performed last. When performing rigid cystoscopy, a 0° degree lens is used for this portion of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following indications for outpatient cystourethroscopy:

  1. Microscopic hematuria or
  2. Voiding dysfunction, or recurrence of urinary incontinence, or
  3. History of recurrent bacterial cystitis
* Age >18
* Patient willingness to enroll
* Patient able to read and understand an English language self- administered questionnaire.

Exclusion Criteria:

* Severe detrussor overactivity
* Interstitial cystitis or chronic urethral or bladder pain
* Acute urinary tract infection
* Urinary retention defined as a post void residual >120cc
* Pregnancy or planning pregnancy within the next 3 months
* Prior urethral surgery
* Dementia or inability to complete questionnaires

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lieschen H Quiroz, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flexible Cystoscopy | Rigid Cystoscopy
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flexible Cystoscopy | Rigid Cystoscopy | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (13.9) | 61.9 (14.8) | 59.7 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race [Count of Participants; unit: Participants]
  Caucasian | 47 | 44 | 91
  Other | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Post Procedural Complications, Including Frequency, Urgency, Infection and Time to Resolution of These Symptoms Between the Two Procedures.
Description: Post procedural complications, including frequency, urgency, infection and time to resolution of these symptoms between the two procedures. Patients were asked to report frequency or urgency as a "yes" or "no"
Time Frame: 1 week after procedure
Population: A total of 42 participants and 43 participants were analyzed from each group, respectively. Some participants may have reported multiple symptoms, which is why the numbers below may exceed to total number of participants analyzed.
Measure: Number; unit: participants
Arm/Group | Rigid Cystoscopy | Flexible Cystoscopy
Number analyzed (Participants) | 42 | 43
participants
  No new symptoms | 17 | 15
  Frequency | 5 | 15
  Urgency | 6 | 11
  Blood in urine | 1 | 0
  Burning with urination | 13 | 14
  Urinary infection | 0 | 0
  Other | 3 | 2

2. Primary Outcome: Duration of Post-procedure Complications
Description: Duration of post-procedure complications, surveyed 1 week post procedure
Time Frame: 1 week after procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Rigid Cystoscopy | Flexible Cystoscopy
Number analyzed (Participants) | 50 | 50
minutes | 5.7 (3.4) | 4.6 (1.8)

3. Secondary Outcome: Visual Analog Pain Scale
Description: The Visual analog pain scale measures patient-reported pain levels from 0-10, with 0 being no pain reported and 10 being the highest level of pain reported. In this study, researchers compared pain levels between females who had rigid and flexible cystoscopies.
Time Frame: Immediately after procedure
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Flexible Cystoscopy | Rigid Cystoscopy
Number analyzed (Participants) | 50 | 50
units on a scale | 0.9 [0.1 to 2.72] | 0.5 [0 to 2.4]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Flexible Cystoscopy | Rigid Cystoscopy
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes